CLINICAL TRIAL: NCT06381206
Title: The Use of Selective Alpha Blockers (Silodosin) in Management of Lower Ureteral Stones Larger Than 6 mm in Diameter
Brief Title: Silodosin in Management of Lower Ureteral Stones
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Diaa Haj Ali, medical doctor Diaa Haj Ali, Syrian Private University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No 475
Record Dates: First submitted 2024-02-09; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Stone, Kidney
Keywords: Silodosin; Lower Ureteral; Ureteral Stones
MeSH Terms: conditions — Kidney Calculi | interventions — silodosin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- case group (Experimental): patients who had given silodosin
  Interventions: Drug: Silodosin
- Control group (No Intervention): patients who had not given silodosin

INTERVENTIONS:
Drug: Silodosin — Selective Alpha Blocker drug
  Arms: case group

SUMMARY:
This research aims to study the effectiveness of silodosin in the management of lower ureter stones larger than 6 mm in diameter in terms of affected ureter (right or left), the size of the stone, the degree of hydronephrosis, the rate of stone expulsion(day), whether the stone was completely expelled or not, and the side effects of silodosin.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the urology Clinic with a distal unilateral ureteral stone larger than 6 mm in diameter.

Exclusion Criteria:

* Patients under 18 years of age
* Pregnant women
* Patients with whom we were unable to contact
* Patients treated with silodosin for another reason
* Single kidney patients
* Patients with bilateral ureter stones
* Patients with deteriorating kidney function
* Patients with grades 3rd and 4th of hydronephrosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Stone expulsion (yes) | 1 year
  patients who were able to expel the stone
Stone expulsion (no) | 1 year
  patients who were not able to expel the stone

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus university, Damascus, Syria